CLINICAL TRIAL: NCT06564779
Title: Development, Standardisation and Standardisation Project for a New Memory Assessment
Acronym: NEM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR240067-NEM
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Memory Disorders
Keywords: Alzheimer; Episodic memory
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group intervention: patients benefiting from the new memory assessment
  Interventions: Other: New memory assessment

INTERVENTIONS:
Other: New memory assessment — The intervention is part of the neuropsychological assessment carried out as part of routine care. It consists of carrying out the neuropsychological tests traditionally used to investigate the diagnostic hypothesis of Alzheimer's disease.

SUMMARY:
Episodic memory (EM) is a neuropsychological marker of Alzheimer's disease (AD) (Thomas-Anterion, 2006). Current tests for its assessment do not take into account the identity and emotional aspects of memory (Van der Linden et al., 2018). However, there are models that integrate links with identity, self-awareness and experience. Pause et al. (2013) propose criteria to create ecological tools, including consideration of the emotional valence of memories and the spatio-temporal context of acquisition. In line with these criteria, we have developed a new tool: the NEM (New evaluation of Episodic Memory). Preliminary studies show different response profiles on the NEM among patients (Launay et al., 2023). We now want to evaluate the relevance of this tool in the differential diagnosis of AD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Ability to understand judged sufficient by the assessor;
* Amnesic MCI profile (Petersen, 2003) during the 1st medical consultation prior to the assessment being prescribed.

Exclusion Criteria:

* Severe auditory and/or visual sensory impairment not compatible with neuropsychological assessment;
* Judged fit to take the test by the assessor;
* Patient under guardianship, curatorship or family guardianship;
* Opposition to data processing.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient attending a memory consultation for suspected Alzheimer's disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Score total NEM (new memory assessment) | baseline
  Sum of the episodic elements

SECONDARY OUTCOMES:
NEM sub-scores | baseline
  Sum of the episodic elements by category
Total RL/RI 16 Recall | baseline
  (Van der Linden et al., 2014)
Delayed Mem Logic Recall | baseline
  (MEM IV, Wechsler, 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Alix LAUNAY, Principal Investigator — Tours University Hospital
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided